CLINICAL TRIAL: NCT02987257
Title: NATIENS: A Phase III Randomized Double-Blinded Placebo Controlled Study to Determine the Optimal Management and Mechanisms of Stevens-Johnson Syndrome and Toxic Epidermal Necrolysis
Brief Title: NATIENS: Optimal Management and Mechanisms of SJS/TEN
Acronym: NATIENS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Ottawa (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Elizabeth J Phillips, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 212370
Record Dates: First submitted 2016-11-25; First posted 2016-12-08 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stevens-Johnson Syndrome; Toxic Epidermal Necrolyses
Keywords: Therapeutics; Management; Etanercept; Supportive Care; Immunopathogenesis; Genetics; Adverse Drug Reaction
MeSH Terms: conditions — Stevens-Johnson Syndrome; Drug-Related Side Effects and Adverse Reactions | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Harmonized supportive care (Placebo Comparator): Harmonized supportive care with etanercept placebo days 1 and 4
  Interventions: Drug: Harmonized supportive care
- Etanercept 50mg sc day 1 and day 4 (Active Comparator): Harmonized supportive care with placebo days 1 and 4
  Interventions: Drug: Harmonized supportive care; Drug: Etanercept 50 mg sc day 1 and day 4

INTERVENTIONS:
Drug: Harmonized supportive care — Harmonized supportive care with and etanercept placebo days 1 and 4
Drug: Etanercept 50 mg sc day 1 and day 4 — Harmonized supportive care with placebo
  Arms: Etanercept 50mg sc day 1 and day 4

SUMMARY:
The North American Therapeutics in Epidermal Necrolysis Syndrome (NATIENS) study is a multicenter double-blind randomized controlled assessment of two arms - one of systemic immunomodulatory therapy (etanercept) and one of supportive care deemed to be the current standard of care. We will leverage the opportunity of this controlled design to collect multiples samples with an aim to discover new genetic and biological markers for prevention and early diagnosis and define cellular and molecular mechanisms to facilitate discovery of promising treatment strategies. This study has been preceded by a planning phase to ensure testing and development of harmonized supportive care infrastructure and operating procedures across sites.

DETAILED DESCRIPTION:
The scientific rationale for this study is the lack of evidence-based treatment for SJS/TEN. The study will aim to establish the most clinically effective therapy for SJS/TEN, as there is currently no level 1A evidence for any treatment above aggressive supportive care which still has equipoise as the standard of care. A multi-centered, two-arm allocated 1:1, double-blind randomized controlled trial with a planned enrollment of 150 patients over 4 years will be undertaken to evaluate which of supportive care or etanercept leads to the shortest time to complete reepithelialization which is the primary outcome. The controlled setting of the clinical trial provides the basis for which samples can be sequentially collected to answer important mechanistic questions. Samples collected during the study will include DNA, PBMC, RNA, plasma, serum, blister fluid cells and supernatant, sloughed epidermis and punch biopsies of skin. Samples will be bio-banked to do immediate targeted high-resolution HLA sequencing, cytokine profiling and single cell multidimensional analyses to identify biological markers that have the potential to predict risk and outcome of SJS/TEN. A population pharmacokinetic study to assess the disposition of etanercept will be done by collecting five samples over the course of the study. Samples will be biobanked for later analysis for other transcriptomic, proteomic whole genome studies. These mechanistic studies will allow us to gain important insights into the immunopathogenesis of SJS/TEN. Our study will be the first to examine in a blinded randomized controlled design both management and mechanisms of SJS/TEN. We anticipate that this will lead to new ways to prevent, diagnosis and treat SJS/TEN, and will create a roadmap and evidence-base for studies in serious immunologically mediated adverse drug reactions and other immunologically mediated diseases.

This protocol represents the only appropriately powered randomized, double-blind mechanistic clinical trial examining therapeutic interventions for SJS/TEN. It will address several significant gaps in knowledge. From a management perspective, it will provide the highest level of supportive care and prove or refute the benefits of etanercept that is a promising therapy for SJS/TEN. The NATIENS trial will also define the standard for systematically assessing the benefit of a systemic intervention for SJS/TEN in prospective studies. We also hope to identify key biomarkers as well as immunologic and genetic determinants for risk, rapid diagnosis, baseline pathophysiology, and mechanisms of response to therapy. The population pharmacokinetics of etanercept will be established for the first time in this critically ill population to improve future dosing strategies and make recommendations. Finally, the protocols and procedures related to patient care will establish a standard for harmonization of care for these patients to provide the best outcomes possible. The study is likely to result in paradigm shifting knowledge regarding SJS/TEN treatment, diagnosis, prevention, and pathogenesis that will lead to improved care for future SJS/TEN patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Subject and/or legally authorized representative must be able to understand and provide informed consent.
3. Erythematous to dusky macules that show evidence of coalescing and/or denuding skin or blistering in a predominantly truncal distribution (Nikolsky sign = sloughing with direct lateral pressure on non-blistered but involved skin should be considered as a supportive feature
4. At least two of the following:

   1. Mucous membrane involvement
   2. Prodromal symptoms including fever, myalgia, and headache
   3. Evidence of disease progression with an increasing number of skin lesions
5. History of a newly used medication within the last 2 months that has not been tolerated for longer than 12 weeks in the past
6. Females of childbearing potential must have a negative pregnancy test prior to randomization.

Exclusion Criteria:

1. Subject or legally authorized representative is not willing to provide informed consent.
2. A serious drug reaction or possible alternative dermatologic diagnosis at the time of initial evaluation not in keeping with drug-induced SJS/TEN (e.g. graft versus host disease).
3. If greater than 5 days has elapsed from onset of initial cutaneous or mucosal signs of the disease as obtained by patient history or documentation.
4. Patients who have received etanercept in the last 6 months.
5. Patients who in time since onset of SJS/TEN illness have received intravenous immune globulin (IVIg) or > 2 doses of pulsed corticosteroid (defined by > 250 mg prednisone equivalent) prior to enrollment in the study.
6. End-stage liver disease (Child Pugh A, B or C or severe liver dysfunction).
7. Grade 2 or higher liver dysfunction (alanine aminotransferase >3 fold or bilirubin >3 fold the upper limit of normal).
8. Any organ transplant.
9. Pre-existing Class III/IV Heart Failure (New York Heart Association Functional Classification).
10. Multiple Sclerosis or other demyelinating diseases.
11. Pregnancy or breastfeeding.
12. Current or past history of immune checkpoint inhibitor therapy for cancer.
13. Absolute need for a drug that interacts with cyclosporine without an appropriate substitution.
14. History of other immunosuppressive or immunomodulatory therapy that could significant impact treatment or interpretation of response to treatment (i.e. azathioprine, methotrexate, mycophenolate mofetil, mycophenolate sodium, rituximab, JAK inhibitors, IL-17 inhibitors, IL-23 inhibitors, other TNF alpha antagonists (see MOP).
15. Use of surgical debridement and/or xenograft.
16. Known positive SARS-CoV-2 on RT-PCR within 10 days prior to screening or within 5 days of admission or symptomatic COVID-19 infection at screening. Symptomatic patients with a positive SARS-CoV-2 on RT-PCR or comparable assay beyond 10 days must be evaluated by the Independent Protocol Monitor.
17. Clinical or radiographic evidence of active tuberculosis or endemic mycoses.
18. History or evidence of any other clinically significant medical or psychiatric disorder, condition or disease that in the opinion of the treating physician would pose a risk or interfere with evaluation or completion of the study such as known sepsis/systemic infection requiring antibiotic therapy.
19. Known hypersensitivity to Enbrel® (etanercept).
20. Receipt of a live attenuated vaccine within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Time to complete re-epithelialization | up to 4 weeks
  Patients will be assessed by two independent raters (burn surgeons, dermatologists, wound care experts) to determine the day of full re-epithelialization. For disagreements on the day of re-epithelialization the case with supporting photographs will be referred to an independent adjudication committee comprised of a minimum of three experts (a burn surgeon, dermatologist, wound care expert). In the instance of death will be the maximum period of re-epithelialization (21 days + 1)

SECONDARY OUTCOMES:
Time to halting of progression of SJS/TEN skin disease | up to 4 weeks
  Progression will be considered significant if there are any new blistering lesions or any new detached or detachable skin.
Mortality | up to 1 year
  Number of participants with mortality at 30 days, 3 months and 1 year
Mortality | up to 4 weeks
  Number of participants with Actual mortality versus expected mortality for each SCORTEN risk
Ocular involvement | up to 1 year or study outcome
  Time to cessation of acute ocular involvement acutely then extent of ocular involvement at follow-up will be assessed by two independent ophthalmology experts. Will be tracked by photography
Infections | up to 4 weeks
  Incidence of nosocomial infections
Hospital length of stay | up to 4 weeks
  Duration of time in hospital
Proportion of patients with Adverse events due to assigned treatment arm | up to 4 weeks
  Adverse events due to assigned treatment arm

OTHER OUTCOMES:
Granulysin, IL-15 and other cytokine measurements | up to 1 year or study outcome
  Featured exploratory secondary outcome measuring difference overtime within an individual as well as differences between treatment arms at various time measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Phillips, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (14):
- United States (14):
  - Valleywise Health Medical Center, Phoenix, Arizona
  - University of California, Davis Medical Center, Sacramento, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Health Burn Center, Gainesville, Florida
  - University of Miami, Ryder Trauma Center, Miami, Florida
  - Emory University at Grady Memorial Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - University of Tennessee Health Sciences Center, Memphis, Tennessee
  - Vanderblt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington, Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data available to other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT02987257/ICF_000.pdf